CLINICAL TRIAL: NCT01141725
Title: Safety and Clinical Activity of Treanda® (Bendamustine HCL) and Idarubicin in Combination Therapy for Patients Age >= 50 With Previously Untreated Acute Myeloid Leukemia and High Risk Myelodysplastic Syndrome
Brief Title: Bendamustine and Idarubicin in Treating Older Patients With Previously Untreated AML or MDS
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2413.00; NCI-2010-01253 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); K12CA076930 (NIH)
Record Dates: First submitted 2010-06-09; First posted 2010-06-10 (Estimated); Results first posted 2017-08-18 (Actual); Last update posted 2017-08-18 (Actual); Status verified 2017-07

CONDITIONS: Adult Acute Myeloid Leukemia With 11q23 (MLL) Abnormalities; Adult Acute Myeloid Leukemia With Del(5q); Adult Acute Myeloid Leukemia With Inv(16)(p13;q22); Adult Acute Myeloid Leukemia With t(15;17)(q22;q12); Adult Acute Myeloid Leukemia With t(16;16)(p13;q22); Adult Acute Myeloid Leukemia With t(8;21)(q22;q22); de Novo Myelodysplastic Syndromes; Myelodysplastic Syndrome With Isolated Del(5q); Untreated Adult Acute Myeloid Leukemia
MeSH Terms: conditions — Congenital Abnormalities; Chromosome 5q Deletion Syndrome | interventions — Bendamustine Hydrochloride; Idarubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (combination chemotherapy) (Experimental): Patients receive bendamustine hydrochloride IV on days 1-5 and idarubicin IV on days 1 and 2. Treatment repeats every 28 days for up to 3 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: bendamustine hydrochloride; Drug: idarubicin

INTERVENTIONS:
Drug: bendamustine hydrochloride — Given IV
  Other Names: bendamustin hydrochloride; bendamustine; cytostasan hydrochloride; Treanda
Drug: idarubicin — Given IV
  Other Names: 4-demethoxydaunorubicin; 4-DMDR; DMDR; IDA

SUMMARY:
This phase I/II trial is studying the side effects and best dose of bendamustine hydrochloride when given together with idarubicin in treating older patients with previously untreated acute myeloid leukemia (AML) or myelodysplastic syndrome (MDS). Drugs used in chemotherapy, such as bendamustine hydrochloride or idarubicin, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Giving more than one drug (combination chemotherapy) may kill more cancer cells

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. The maximum tolerated dose (MTD) that is associated with a complete remission (CR) rate of at least 40%, and a rate of grade 3-4 extramedullary toxicity < 30% in patients aged 50 or older with previously untreated AML or high-risk MDS.

SECONDARY OBJECTIVES:

I. The disease-free survival (DFS), and overall survival (OS) after therapy at each level of the dosing strategy.

OUTLINE: This is a phase I, dose-escalation study of bendamustine hydrochloride followed by a phase II study.

Patients receive bendamustine hydrochloride intravenously (IV) on days 1-5 and idarubicin IV on days 1 and 2. Treatment repeats every 28 days for up to 3 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months for 2 years and then annually thereafter for 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of untreated AML or MDS with 10-19% marrow blasts; patients may be enrolled if they received prior treatment with demethylating agents specifically for the purpose of treating MDS or if they have received a single dose of cytarabine for the control of symptoms related to AML
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0-2
* Serum creatinine =< 2.0 mg/dL; if serum creatinine > 2.0 mg/dL, then the estimated glomerular filtration rate (GFR) must be > 50 mL/min/1.73 m^2 as calculated by the Modification of Diet in Renal Disease equation
* Serum bilirubin =< 1.5 x upper limit of normal (ULN)
* Aspartate transaminase (AST)/alanine transaminase (ALT) =< 2.5 x ULN
* Alkaline phosphatase =< 2.5 x ULN
* Capable of understanding the investigational nature, potential risks and benefits of the study, and able to provide valid informed consent
* Males should be willing to use an effective contraceptive method during the study and for a minimum of 6 months after study treatment
* Women must be postmenopausal or must be willing to use an acceptable method of contraception to avoid pregnancy for the entire period of the study and for at least 3 months after the study; a postmenopausal woman is defined as a woman who has experienced amenorrhea > 12 consecutive months or a woman on hormone replacement therapy with documented follicle-stimulating hormone (FSH) level > 35 mIU/mL; for patients in whom menopausal state is in question, a negative pregnancy test will be required prior to enrollment

Exclusion Criteria:

* Current concomitant chemotherapy, radiation therapy, or immunotherapy other than as specified in the protocol
* Use of investigational agents within 30 days or any anticancer therapy within 2 weeks before study entry with the exception of hydroxyurea or single-dose cytarabine; subjects who are enrolled with high risk MDS (specifically) may have prior treatment with drugs in the class called "demethylating agents"; examples of these drugs include 5-azacytidine (azacitidine) and 5-azadeoxycytidine (decitabine), and may include approved or experimental drugs not currently used, which fall into this class and may be developed in the future; the patient must have recovered from all acute toxicities from any previous therapy
* Have any other severe concurrent disease, or have a history of serious organ dysfunction or disease involving the heart, kidney, liver, or other organ system that may place the patient at undue risk to undergo treatment
* Patients with a systemic fungal, bacterial, viral, or other infection not controlled (defined as exhibiting ongoing signs/symptoms related to the infection and without improvement, despite appropriate antibiotics or other treatment)
* Pregnant or lactating patients
* Any significant concurrent disease, illness, or psychiatric disorder that would compromise patient safety or compliance, interfere with consent, study participation, follow up, or interpretation of study results
* Known hypersensitivity to bendamustine (bendamustine hydrochloride) or idarubicin
* Clinical evidence suggestive of central nervous system (CNS) involvement with leukemia unless a lumbar puncture confirms the absence of leukemic blasts in the cerebrospinal fluid (CSF)
* Have had a diagnosis of another malignancy, unless the patient has been disease-free for at least 3 years following the completion of curative intent therapy
* Other circumstances in which patients with prior malignancies are not excluded, include the following:

  * Patients with treated non-melanoma skin cancer, in situ carcinoma, or cervical intraepithelial neoplasia, regardless of the disease-free duration, if definitive treatment for the condition has been completed
  * Patients with organ-confined prostate cancer with no evidence of recurrent or progressive disease based on prostate-specific antigen (PSA) values if hormonal therapy has been initiated, or a radical prostatectomy or definitive radiotherapy has been performed
  * Concurrent hormonal therapy is allowed

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2010-09; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Pagel, Principal Investigator — Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium
Locations (1):
- Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium, Seattle, Washington, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Bendamustine Dose of 45mg/m2/Day: Patients receive bendamustine hydrochloride 45mg/m2 IV on days 1-5 and idarubicin 12mg/m2 IV on days 1 and 2.
  Treatment repeats every 28 days for up to 3 courses in the absence of disease progression or unacceptable toxicity.
- Bendamustine Dose of 60mg/m2/Day: Patients receive bendamustine hydrochloride 60mg/m2 IV on days 1-5 and idarubicin 12mg/m2 IV on days 1 and 2.
  Treatment repeats every 28 days for up to 3 courses in the absence of disease progression or unacceptable toxicity.
- Bendamustine Dose of 75mg/m2/Day: Patients receive bendamustine hydrochloride 75mg/m2 IV on days 1-5 and idarubicin 12mg/m2 IV on days 1 and 2.
  Treatment repeats every 28 days for up to 3 courses in the absence of disease progression or unacceptable toxicity.
Period: Overall Study
Arm/Group | Bendamustine Dose of 45mg/m2/Day | Bendamustine Dose of 60mg/m2/Day | Bendamustine Dose of 75mg/m2/Day
Started | 3 | 33 | 3
Completed | 3 | 33 | 3
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Combination Chemotherapy)
Number analyzed (Participants) | 39
Age, Continuous [Median (Full Range); unit: years] | 73 [56 to 82]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24
  Male | 15
Region of Enrollment [Number; unit: participants]
  United States | 39
ECOG [Count of Participants; unit: Participants] — ECOG performance status
  * grade 0: fully active, able to carry on all pre-disease performance without restriction
  * grade 1 : restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work
  * grade 2 : ambulatory and capable of all selfcare but unable to carry out any work activities, up and about more than 50% of waking hours
  Participants
    ECOG 0 | 0
    ECOG 1 | 35
    ECOG 2 | 4

OUTCOME MEASURES:

1. Primary Outcome: Response
Description: Assessed by cytogenetics/fluorescence in situ hybridization (FISH) and flow cytometry of blood and bone marrow samples. The response criteria defined by Cheson et al. will be used in this study. These criteria are: morphologic leukemia-free state; morphologic complete remission (CR); cytogenetic CR (CRc); molecular CR (CRm); morphologic CR with incomplete blood count recovery (CRi); partial remission (PR); treatment failure; recurrence (progressive disease).
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Groups:
- Treatment A: Patients receive bendamustine hydrochloride 45mg/m2 IV on days 1-5 and idarubicin 12mg/m2 IV on days 1 and 2.
  Treatment repeats every 28 days for up to 3 courses in the absence of disease progression or unacceptable toxicity.
- Treatment B: Patients receive bendamustine hydrochloride 60mg/m2 IV on days 1-5 and idarubicin 12mg/m2 IV on days 1 and 2.
  Treatment repeats every 28 days for up to 3 courses in the absence of disease progression or unacceptable toxicity.
- Treatment C: Patients receive bendamustine hydrochloride 75mg/m2 IV on days 1-5 and idarubicin 12mg/m2 IV on days 1 and 2.
  Treatment repeats every 28 days for up to 3 courses in the absence of disease progression or unacceptable toxicity.
Arm/Group | Treatment A | Treatment B | Treatment C
Number analyzed (Participants) | 3 | 33 | 3
Participants
  CR | 0 | 10 | 1
  CRi | 0 | 2 | 0
  No CR | 3 | 21 | 2

2. Primary Outcome: Incidence of Greater Than or Equal to Grade 3 Toxicity
Description: Toxicities will be graded using the National Cancer Institute (NCI) Common Toxicity Criteria version 3.0.
Time Frame: Up to day +100 after end of therapy or until the patient received an alternative treatment for leukemia, whatever happens earlier
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment A | Treatment B | Treatment C
Number analyzed (Participants) | 3 | 33 | 3
Participants | 0 | 0 | 2

3. Primary Outcome: Maximum Tolerated Dose
Description: A bayesian approach to estimate the MTD of bendamustine associated with a CR rate of at least 40% and with <30% grade 3-4 non-haematological toxicity was used (Wathen et al, 2008).The MTD of bendamustine in combination with idarubicin was determined after two cases of grade 3 toxicity were noted in the three patients entered at the 75 mg/m2 dose. The DLTs were congestive heart failure and mucositis in one patient each. Patients subsequent to this were treated at the 60 mg/m2 bendamustine dose.
Time Frame: 6 months
Measure: Number; unit: mg/m2
Arm/Group | Treatment (Combination Chemotherapy)
Number analyzed (Participants) | 39
mg/m2 | 60

4. Primary Outcome: Median Survival
Description: In a five year following, the median survival was obtained.
Time Frame: 5 years
Measure: Median (Full Range); unit: months
Arm/Group | Treatment (Combination Chemotherapy)
Number analyzed (Participants) | 39
months | 7.2 [1 to 22]

5. Secondary Outcome: Disease-free Survival (DFS)
Description: In a five year following, the disease free survival was obtained.
Time Frame: 5 years
Population: Data for this Outcome Measure was not collected per dose level and is unavailable.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Treatment (Combination Chemotherapy)
Number analyzed (Participants) | 39
days | 235 [83 to 277]

ADVERSE EVENTS:
Time Frame: 6 months
Description: Other (Not Including Serious) Adverse Events were not collected/assessed.
Groups:
- Treatment (Combination Chemotherapy): Patients receive bendamustine hydrochloride IV on days 1-5 and idarubicin IV on days 1 and 2. Treatment repeats every 28 days for up to 3 courses in the absence of disease progression or unacceptable toxicity.
  bendamustine hydrochloride: Given IV
  idarubicin: Given IV
  Adverse event report was not collected by dose level.
Arm/Group | Treatment (Combination Chemotherapy)
All-Cause Mortality (participants affected / at risk) | 4/39
Serious Adverse Events (participants affected / at risk) | 29/39
Other Adverse Events (participants affected / at risk) | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Combination Chemotherapy) (N=39)
Febrile Neutropenia (Blood and lymphatic system disorders) | 29 (29)
Fungal infection (Infections and infestations) | 4 (4)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Cellulitis (Skin and subcutaneous tissue disorders) | 2 (2)
Bacteraemia (Infections and infestations) | 2 (2)
Sepsis (Infections and infestations) | 2 (2)
Sinusitis (Infections and infestations) | 1 (1)
Platelet transfusion refractory (Blood and lymphatic system disorders) | 1 (1)
Heart Failure (Cardiac disorders) | 1 (1)
Atrial Fibrillation (Cardiac disorders) | 1 (1)
Severe mucositis (Infections and infestations) | 1 (1)
Intracranial bleeding (Blood and lymphatic system disorders) | 1 (1)
Clostridium difficile infection (Infections and infestations) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dehydration (General disorders) | 1 (1)
Acute renal injury (Renal and urinary disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No